CLINICAL TRIAL: NCT05171972
Title: Assessing Reduced Oligodendrocyte-specific Cytotoxicity of Peripheral Blood Leukocytes in Patients With Multiple Sclerosis Following Treatment With Ofatumumab
Brief Title: Reduced Oligodendrocyte-specific Cytotoxicity and Ofatumumab Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Brett T. Lund, Associate Professor of Research, University of Southern California
Other Study IDs: HS-21-00540
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Kesimpta; Ofatumumab
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Relapsing-remitting Multiple Sclerosis: Enrolled subjects in this group will have clinically definite Multiple Sclerosis as defined by the revised McDonald criteria of the relapsing-remitting form with an Expanded Disability Status Scale (EDSS) score of 0 to 5.5 and will be treated with Ofatumumab.
  Interventions: Drug: Ofatumumab
- Healthy Control Subjects: Enrolled subjects must not have clinically definite Multiple Sclerosis as defined by the revised McDonald criteria, any other autoimmune disease, demyelinating co-morbidity, neurological disease or immune system altering disease.

INTERVENTIONS:
Drug: Ofatumumab — This investigator-initiated study will be carried out secondary to the discussion of treatment with Ofatumumab and thus our study will not influence or impact the determination of the suitability for candidates to commence therapy with Ofatumumab. This decision will be made by the patient's physician as part of the patient's standard care, and will occur independently of this study. Patients to be enrolled in this longitudinal study will only be asked if they would like to take part if their clinician independently chooses Ofatumumab as a treatment option.
  Other Names: Kesimpta
  Groups: Relapsing-remitting Multiple Sclerosis

SUMMARY:
In this study the investigators wish to test the hypothesis that the repertoire of solutes secreted by leukocytes isolated from patients with relapsing-remitting forms of Multiple Sclerosis (MS) following 6 months of treatment with Ofatumumab (Kesimpta®) will be less toxic to mouse-derived oligodendrocyte lineage cells, grown in a dish, than solutes secreted by the same leukocyte populations prior to treatment with Ofatumumab.

DETAILED DESCRIPTION:
Background and Rationale:

The role of B-cells in multiple sclerosis (MS) pathogenesis is still not fully understood, however studies have shown that: 1) intrathecal synthesis of immunoglobulin can be detected in the cerebral spinal fluid of >90% of MS patients; 2) there are multiple clonally expanded B-cell populations in chronic MS brain lesions; 3) ectopic lymphoid follicles containing proliferating B-cells have been identified within the meninges of secondary progressive MS patients; and 4) anti-B cell depleting therapies have been shown to have clinical benefit in MS. In addition to these findings B-cells have been shown to:

* Secrete autoantibodies.
* Serve as antigen-presenting cells.
* Facilitate T-cell activation.
* Contribute to the micro-environment by local secretion of immune mediators such as cytokines and chemokines.

It is important that investigators not only understand the clinical effects of B-cell depletion, but also, critically, that investigators understand the ongoing mechanisms of action following treatment with Ofatumumab. Specifically, how the remaining pathogenic leukocyte populations, such as T-cells, monocytes, neutrophils and natural killer (NK) cells are modulated indirectly by Ofatumumab such that they may be less pathogenic to the myelinating oligodendrocyte population.

Ofatumumab is an anti-CD20 human monoclonal antibody that has demonstrated efficacy in lowering relapse rates, magnetic resonance Imaging (MRI) activity and neurofilament light (NF-L) levels, as well as significant reductions in confirmed disability worsening in patients with relapsing forms MS.

The exact role(s) of B cells in MS pathogenesis are still unclear at present, as are the events that lead to oligodendrocyte death and dysfunction. Oligodendrocytes are the myelinating cells of the central nervous system (CNS), and demyelination and oligodendrocyte death are critical events in the disease process of MS. At present no current approved MS drug therapies are targeted to directly protecting against oligodendrocyte loss and dysfunction or aimed at enhancing repair of the CNS. The proposed studies in this application are novel in that effect(s) of Ofatumumab treatment in MS has not been previously studied in oligodendrocyte or oligodendrocyte progenitor cell (OPC) populations. The outcomes from this study could identify an additional mode of action of Ofatumumab treatment, with effects that could indirectly benefit the CNS.

Specific Aims:

For this study, the investigators propose that the long-term mechanism of action associated with the beneficial clinical outcomes of Ofatumumab therapy in MS is not only due to the direct effect of removing circulating B-cells, but is also due to the subsequent alteration in immune homeostasis with an accompanied reduction in cytotoxic secretory products from leukocyte subsets including T cells, monocytes, neutrophils and NK cells. The study has two specific aims:

For Specific Aim 1 (primary objective) the investigators will determine if solutes secreted by T cells, monocytes, neutrophils or NK cells isolated from patients with relapsing-remitting forms of MS following 6 months (M06) of treatment with Ofatumumab are less toxic to mouse-derived oligodendrocytes and their progeny (OPC) than solutes secreted by the same sub-populations of leukocytes collected prior to treatment (M00 drug naive). In this aim, the primary outcome will be to assess measures of oligodendrocyte and OPC death, and mitochondrial dysfunction.

For Specific Aim 2 (exploratory objective) the investigators will identify the factor(s) responsible for inducing oligodendrocyte and OPC stress (comparing M06 supernatant samples to M00) by firstly using a cytokine array approach followed, if needed, by a 2D-electrophoresis LC-MS proteomic approach. The investigators will also perform additional analyses that will explore altered microglial and astrocyte responses following treatment with solutes secreted from leukocyte sub-populations at M00 and M06 in MS patients.

Study Population:

For this prospective longitudinal study the investigators will recruit 20 patients with clinically definite relapsing-remitting MS (RR-MS) (as defined by the revised McDonald criteria) who will be treated with Ofatumumab (Kesimpta). The investigators will also recruit 20 healthy control (HC) subjects. For these studies, RR-MS patients will serve as their own internal control and the investigators will compare changes over time on Ofatumumab with pre-treatment measures. In addition, RR-MS patient samples will be compared to healthy control leukocyte sub-population supernatants. All RR-MS patients will be prescribed and treated with Ofatumumab as part of their standard of care from their treating provider, with the exception of the HC subjects who receive no treatment.

Procedures and Data Collection:

All RR-MS patients will be selected from those currently being seen by physicians at the Multiple Sclerosis Comprehensive Care Center at University of Southern California (USC) Keck School of Medicine or the LAC+USC Medical Center, Multiple Sclerosis Clinic, and for whom the physician has already deemed Ofatumumab would be a logical treatment alternative. The investigators will not be assessing eligibility for Ofatumumab treatment as criteria for inclusion in this investigator-initiated trial (IIT). The investigators expect enroll subjects over a 10-12 month recruitment phase. The investigators expect the last patient sample to be collected 18 months following commencement of the study with final analysis of data completed 27 months after study commencement. For the Ofatumumab cohort, the investigators will collect ~80ml blood from enrolled patients at M00 (baseline, naive to drug), and will collect a further 80ml of blood at M06 (months 5-6 prior to the 6-month Ofatumumab injection). For the HC cohort, the investigators will collect ~80ml blood from enrolled subjects at only one time point. Blood samples will be processed and leukocyte sub-populations isolated for culture.

ELIGIBILITY:
Inclusion Criteria:

RR-MS patients only:

This investigator-initiated study/trial (IIT) will be carried out secondary to the discussion of treatment with Ofatumumab and thus our study will not influence or impact the determination of the suitability for candidates to commence therapy with Ofatumumab. This decision will be made by the patient's physician as part of the patient's standard care, and will occur independently of this study. Patients to be enrolled in this longitudinal study will only be asked if they would like to take part in this IIT if their clinician independently chooses Ofatumumab as a treatment option:

* Patients must qualify to receive treatment with Ofatumumab (Kesimpta), according to the Multiple Sclerosis Comprehensive Care Center at USC Keck School of Medicine or LAC+USC Medical Center and meet the inclusion criteria defined in, and aligned with, the US Kesimpta (Ofatumumab) Prescribing Information.
* Patients must have clinically definite Multiple Sclerosis as defined by the revised McDonald criteria of the relapsing-remitting form with an Expanded Disability Status Scale (EDSS) score of 0 to 5.5.
* Patients must be treatment naive to Ofatumumab (Kesimpta)
* Patients must have the ability to understand and sign this study-specific IRB-approved informed consent form.
* Patients must be willing to donate ~80ml of blood each for M00 and M06 that will be used for testing the specific aims described in this proposal.
* Patients must have a lymphocyte count within the normal range at baseline (3.8-10.8 x1,000/ml)

Healthy Control Subjects only:

* Patients must not have clinically definite Multiple Sclerosis as defined by the revised McDonald criteria, any other autoimmune disease, demyelinating co-morbidity, neurological disease or immune system altering disease (e.g. HIV).
* Patients must have the ability to understand and sign this study-specific IRB-approved informed consent form.
* Patients must be willing to donate ~80ml of blood at one time only that will be used for testing the specific aims described in this proposal.
* Patients must have a lymphocyte count within the normal range at baseline (3.8-10.8 x1,000/ml).

Exclusion Criteria:

RR-MS patients only:

* Treatment with any of the following within 90 days of commencing treatment with Ofatumumab: teriflunomide (Aubagio®), IV immunoglobulin or plasmapheresis.
* Previous treatment with natalizumab (Tysabri®) within 30 days of commencing treatment with Ofatumumab.
* Documented relapse within 30 days prior to baseline.
* Systemic corticosteroid therapy within 4 weeks prior to baseline.
* Prior treatment with Mitoxantrone, Cyclophosphamide, Cyclosporine, Azathioprine or Methotrexate or any other immunosuppressant, or total body irradiation or bone marrow transplantation.
* Prior treatment with a B-cell targeted therapies (e.g., rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab).
* Prior treatment with alemtuzumab (Lemtrada®).
* Current supplemental treatment with high dose biotin.
* Women who are pregnant, lactating, breast feeding or of childbearing age who do not consent to approved contraceptive use during the study.
* Prior or current treatment with a drug that is experimental
* Meet any of the exclusion criteria defined in, and aligned with, the US Kesimpta/Ofatumumab Prescribing Information.

Healthy Control Subjects:

* Treatment with any FDA-approved drug or experimental drug for any condition.
* Systemic corticosteroid therapy within 4 weeks prior to blood collection.
* Women who are pregnant, lactating, or could be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this prospective longitudinal study the investigators will recruit 20 patients with clinically definite relapsing-remitting MS (as defined by the revised McDonald criteria) who will be treated with Ofatumumab (Kesimpta). Patients will be recruited from the Multiple Sclerosis Comprehensive Care Center at USC Keck School of Medicine and the LAC+USC Medical Center, Multiple Sclerosis Clinic. The investigators will also recruit 20 healthy control (HC) subjects. Healthy controls will be age and sex matched to the RR-MS population as much as possible.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-29 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of oligodendrocyte death and mitochondrial dysfunction comparing supernatant samples from patients after 6 months treatment (M06) to pre-treatment, drug naïve supernatants (M00) and to supernatants collected from healthy control subjects | 27 months
  To determine if solutes secreted by T cells, monocytes, neutrophils or NK cells isolated from patients with relapsing-remitting forms of MS following 6 months (M06) of treatment with Ofatumumab are less toxic to mouse-derived oligodendrocytes and their progeny (OPC) than solutes secreted by the same sub-populations of leukocytes collected prior to treatment (M00 drug naive), and how this compares to samples from healthy control subjects.

SECONDARY OUTCOMES:
Identify factor(s) associated with oligodendrocyte and OPC stress/death | 27 months
  Perform analysis of M06 and M00 supernatant samples to identify factor(s) associated with oligodendrocyte and OPC stress/death. Approaches utilized: 1) Cytokine bead array; 2D-electrophoresis LC-MS proteomic analyses and 3) Examination of altered microglial and astrocyte cell number and morphology in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Eve Kelland, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No